CLINICAL TRIAL: NCT02143739
Title: The Severity of Newly Diagnosed Asthma Patients and the Result of Initial 12 Weeks Treatment in China.
Acronym: INITIAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RCN-XXX-2013/2
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly diagnosed asthma patients: The patient population will be outpatients, men or women, ≥18 years of age, Newly diagnosed asthma patients who are not on inhaled gluococorticosteroid within 3 months.The patient population should not have COPD(chronic obstructive pulmonary diseases) history, or asthma exacerbation.

SUMMARY:
The primary objective of the NIS is to evaluate the severity of newly diagnosed asthma patients based on Global Initiative for Asthma (GINA) severity category (GINA 2006 update).

DETAILED DESCRIPTION:
This is a multi-centre, prospective non-interventional study planned to be conducted in China. The study aims to recruit about 5000 newly diagnosed patients from about 50 tier 3 hospitals with respiratory department. Each site recruits about 50-150 patients.

The primary variable will be distribution of severity based on GINA definition (GINA 2006 update) at baseline in the total population.

There will be 4 visits for this study, Informed consent and following study procedures (ACQ-5(asthma control questionnaire), severity assessment) will be done at visit 1. After that, according to clinical practice in China patients usually go to the clinic every 4 weeks. Asthma control status, ACQ-5 and sever exacerbation will be assessed at each clinic visit till 12 weeks (visit 2, 3, 4).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed asthma patients who are not on inhaled gluococorticosteroid within 3 months.
2. Out-patient with an age of 18 years and above
3. Signed and dated informed consent The prescription of the medicinal product is clearly separated from the decision to include the subject in the NIS. Generally, asthma medication refers to those recommended in GINA guideline (GINA2012 update) and decided by investigator.

Exclusion Criteria:

1. Participating in any clinical trial during the last 90 days
2. Have COPD
3. With asthma exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be outpatients, men or women, ≥18 years of age, Newly diagnosed asthma patients who are not on inhaled gluococorticosteroid within 3 months.The patient population should not have COPD history, or asthma exacerbation.
Sampling Method: Probability Sample
Enrollment: 4817 (Actual)
Dates: Start 2014-06-07 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Asthma Severity assessment based on GINA definition (GINA 2006 update) at baseline in the total population | Day 1
  severity based on GINA definition (GINA 2006 update) at baseline in the total population.

SECONDARY OUTCOMES:
evaluate the control level of initial 12 weeks treatment based on Assessment of Current Clinical Control in GINA (GINA 2012 update). | up to 3 months
  The asthma control status assessment will be based on Assessment of Current Clinical Control in GINA (GINA 2012 update).

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Lin, PhD, Principal Investigator — China-Japan Friendship Hospital
Locations (30):
- China (30):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changshu
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Daping
  - Research Site, Fuzhou
  - Research Site, Guangyuan
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Mianyang
  - Research Site, Nantong
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou

REFERENCES:
- [Background] Lin JT, Chen P, Zhou X, Sun TY, Xie CM, Xiu QY, Yao WZ, Yang L, Yin KS, Zhang YM. Budesonide/formoterol maintenance and reliever therapy in Chinese patients with asthma. Chin Med J (Engl). 2012 Sep;125(17):2994-3001. PMID 22932169
- [Background] Rabe KF, Vermeire PA, Soriano JB, Maier WC. Clinical management of asthma in 1999: the Asthma Insights and Reality in Europe (AIRE) study. Eur Respir J. 2000 Nov;16(5):802-7. doi: 10.1183/09031936.00.16580200. PMID 11153575
- [Background] Thompson PJ, Salvi S, Lin J, Cho YJ, Eng P, Abdul Manap R, Boonsawat W, Hsu JY, Faruqi RA, Moreno-Cantu JJ, Fish JE, Ho JC. Insights, attitudes and perceptions about asthma and its treatment: findings from a multinational survey of patients from 8 Asia-Pacific countries and Hong Kong. Respirology. 2013 Aug;18(6):957-67. doi: 10.1111/resp.12137. PMID 23730953
- [Background] Zhao J; National Parents of Asthmatic Children KAP Project Team. [Asthma control status in children and related factors in 29 cities of China]. Zhonghua Er Ke Za Zhi. 2013 Feb;51(2):90-5. Chinese. PMID 23527968
- [Result] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Result] Juniper EF, O'Byrne PM, Roberts JN. Measuring asthma control in group studies: do we need airway calibre and rescue beta2-agonist use? Respir Med. 2001 May;95(5):319-23. doi: 10.1053/rmed.2001.1034. PMID 11392570
- [Derived] Lin J, Fu X, Jiang P, Song W, Hu X, Jie Z, Liu C, He Z, Zhou X, Tang H. INITIAL - An observational study of disease severity in newly diagnosed asthma patients and initial response following 12 weeks' treatment. Sci Rep. 2019 Feb 4;9(1):1254. doi: 10.1038/s41598-018-36611-w. PMID 30718519
- See also: 10573240 — https://www.ncbi.nlm.nih.gov/pubmed/?term=10573240
- See also: 11392570 — https://www.ncbi.nlm.nih.gov/pubmed/?term=11392570
- See also: 22932169 — https://www.ncbi.nlm.nih.gov/pubmed/?term=22932169
- See also: 11153575 — https://www.ncbi.nlm.nih.gov/pubmed/?term=11153575
- See also: 23730953 — https://www.ncbi.nlm.nih.gov/pubmed/?term=23730953
- See also: 23527968 — https://www.ncbi.nlm.nih.gov/pubmed/?term=23527968
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2991&filename=synopsis-redacted.pdf